CLINICAL TRIAL: NCT03533764
Title: Translating an Evidence-based Urban Asthma Program for Rural Adolescents: Testing Effectiveness & Cost-effectiveness and Understanding Factors Associated With Implementation
Brief Title: Rural Asthma Effectiveness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Medical University of South Carolina (Other); NYU Langone Health (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jean-Marie Bruzzese, Professor of Applied Developmental Psychology (in Nursing), Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AAAR4130; R01HL136753 (NIH)
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Asthma
Keywords: Asthma Self-Management for Adolescents (ASMA); Community Health Workers (CHW)
MeSH Terms: conditions — Asthma | interventions — MUSK protein, human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research assistants who will interview study participants will be blind to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthma Self-Management for Adolescents (Experimental): Asthma Self-Management for Adolescents (ASMA) consists of three complementary components: (1) an 8- week intervention for students; (2) caregiver education; and (3) education for students' medical providers.
  Interventions: Behavioral: ASMA
- Attention Control (No Intervention): In 3 group sessions and 5 one-on-one sessions, held at school during the school day, students will receive information about asthma and other health topics relevant to adolescents (e.g., nutrition, safety). They will learn to monitor their health by using diaries to record behaviors, such as what they eat, and/or their sleep patterns. Students will be referred to their medical providers for asthma and other health concerns; if they do not have a provider, they are given referrals in their community.

INTERVENTIONS:
Behavioral: ASMA — ASMA, grounded in social cognitive theory and utilizing motivational interviewing techniques, guides adolescents in their transition to being consumers and teaching them to navigate the health system, including overcoming challenges to health care access. Briefly, it consists of three complementary components: (1) an 8- week intervention for students; (2) caregiver education; and (3) education for students' medical providers.
  Arms: Asthma Self-Management for Adolescents

SUMMARY:
The investigators will test if their intervention, Asthma Self-Management for Adolescents (ASMA), an 8-week, high school-based intervention for teenagers, improves asthma in rural high school students with uncontrolled asthma when delivered by CHWs. The investigators will also test the cost-effectiveness of ASMA, and examine the barriers and facilitators of ASMA's widespread implementation.

DETAILED DESCRIPTION:
Asthma, the most common pediatric chronic illness, has high prevalence and morbidity among adolescents. Despite this, there are few interventions for high school students, and none have been tested when delivered by Community Health Workers (CHWs) or in rural areas. This represents a significant limitation because the CHW model has been shown to be successful in clinic- and home-based interventions. Also, rural adolescents with asthma represent a very large population. Given the high prevalence of asthma in this group, this oversight is a significant public health concern. Cost effectiveness analyses and implementation research are also lacking in asthma intervention research. This study addresses these treatment and methodological gaps. The investigators developed and established the efficacy of Asthma Self-Management for Adolescents (ASMA), an 8-week, high school-based intervention, in urban Hispanic and African American adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents who are at least 13.0 at the time of consent
* Teenager reports having a prior asthma diagnosis, and in the last 12 months has: (a) used prescribed asthma medication and (b) uncontrolled asthma, defined as: (i) symptoms 3+ days a week; (ii) night awakenings 3+ nights per month; (iii) 2+ ED visits; or (iv) 1+ hospitalization for asthma; and
* Adolescents are English proficient

Exclusion Criteria:

• Co-morbid diseases that affect lung functioning.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Number of night awakenings due to asthma symptoms | Up to 1 year
  Teens and caregivers report the frequency of night awakenings in the prior weeks.
Number of days with asthma-related activity limitations | Up to 1 year
  Teens and caregivers report the frequency of limitations due to asthma in the prior weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Bruzzese, PhD, Principal Investigator — Columbia University
Locations (1):
- Medical University of South Carolina (MUSC), Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All data shared between sites will be de-identified by HIPAA standards using the "safe-harbor" method (i.e., all 18 identifiers will be stripped) prior to being scanned and stored on a password-protected webserver.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available for up to 7 years from the end of the study.
Access Criteria: Deidentified data.